CLINICAL TRIAL: NCT06853639
Title: Analysis of Oral Health of Students and Former Students of Undergraduate and Postgraduate Programs at the University of São Paulo: A Cohort Study
Brief Title: Analysis of Oral Health of Students and Former Students of Undergraduate and Postgraduate Programs at the University of São Paulo.
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Giuseppe Alexandre Romito, Head of Periodontics Division, University of Sao Paulo
Other Study IDs: FOUSP Cohort study
Record Dates: First submitted 2025-02-17; First posted 2025-03-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Oral Health
Keywords: oral health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dental students: Dental students: people who are aware of oral health problems and adhere to ideal means of prevention.
- Non-Dental students: Non-dental students: people who have little awareness of oral health problems and have unknown adherence to ideal means of prevention.

SUMMARY:
This study aims to evaluate oral and systemic health conditions among students and former students of undergraduate and postgraduate programs at the University of São Paulo over five years. The primary focus is to understand how oral health impacts academic performance and attendance, providing insights for health promotion strategies within the university community.

DETAILED DESCRIPTION:
The study employs a prospective cohort design to explore multiple health-related outcomes, including periodontal health, oral health literacy, and the prevalence of caries. The data collected will also examine social and behavioral predictors of oral health, such as dietary habits, stress, and use of substances like tobacco and electronic cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Current and former undergraduate and postgraduate students of the University of São Paulo.

Exclusion Criteria:

* 1. Individuals who do not consent to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Undergraduate and graduate students at the University of São Paulo
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
Plaque index | through study completion, an average of 5 years
  Primary outcome: plaque index

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe A Romito, Principal Investigator — University of Sao Paulo
Locations (1):
- Faculdade de Odontologia da USP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided